CLINICAL TRIAL: NCT03568825
Title: Randomized Two-dimensional Between-patient Response Surface Pathway Design With Two Interventional- and One Response Variable in Estimating Minimum Efficacy Dose of Osteopathic Manual Therapy in Treatment of Gastroesophageal Reflux Disease
Brief Title: Response Surface Pathway Design With Two Interventional- and One Response Variable in Estimating Minimum Efficacy Dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Meddoc (Other)
Responsible Party: Principal Investigator, Prof Stig Larsen, Professor, Meddoc
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GERD_III_2016-936
Record Dates: First submitted 2018-06-13; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: GERD
Keywords: Two-dimensional randomized response surface pathway design; Osteopathic Manual Therapy; OMT in treatment of GERD; Dose-response
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: The study is a RSP designed multicenter study with two interventional- and one response variable. The two-interventional variable were Number of OMTs and Interval in days between each treatment. The GERD variables were degrees of Heartburn, Chest pain, Acid in mouth, Epigastric pain and "Thoracic pain". The response variable were percent reduction in sum of the GERD variables from baseline in 4 categories. Each of the two RSP designs consisted of three dose levels. Three GERD patients were allocated to the first design level given six OMT with five days' interval. Based on the results obtained from the first design level, five patients were subsequently included to the second design level. The number of OMT's and interval between each treatment was separately determined. Seven patients were included to the third design level and given number of OMT's and interval between treatments calculated based on results obtained from the second design level.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Number of Osteopatic Manual Therapy (Experimental): Intervention: OMT. Osteopatic Manual treatment consisting of Thoracic spine, Diaphragm mobilisation, Traction of the cardia and posture correction.
  Interventions: Procedure: Osteopatic Manual Therapy (OMT)
- Interval in days between each OMT (Experimental): Intervention: OMT. The time between each OMT's is calculated by the study design. Each OMT intervantion consists of Thoracic spine and Diaphragm mobilisation, Traction of the cardia and Posture correction.
  Interventions: Procedure: Osteopatic Manual Therapy (OMT)

INTERVENTIONS:
Procedure: Osteopatic Manual Therapy (OMT) — OMT consisting of following interventions; thoracic spine and diaphragm mobilisation, traction of the cardia and posture correction.

SUMMARY:
Response Surface Pathway (RSP) design was previously developed for dose-finding studies with one interventional and one response variable, but RSP to higher dimensions is requested. The aim of this study is to introduce and evaluate the RSP design with two interventional and one response variable exemplified by estimating Minimum Efficacy Dose (MED) of Osteopathic Manual Therapy (OMT) in treatment of gastroesophageal reflux disease (GERD).

DETAILED DESCRIPTION:
15 GERD patients, divided in three design-level with three, five and seven patients. The study was performed as a two-dimensional randomized, between-patient RSP designed multicenter study with two interventional- and one response variable. The interventional variables "Number of OMT's" and "Treatment Interval" with common response variable formed two independent one-dimensional randomized between-patient RSP studies. The response variable was the percent reduction in sum of the five GERD score from baseline. Three GERD patients were allocated on the first design level given six OMT with five days' interval. Based on results obtained in the first and second design level, five patients were included to the second design level and seven to the third.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosed Gastroesophigual Reflux Disease
* Known effect of anti-reflux medication

Exclusion Criteria:

* Hiatus hernia ≥5 cm
* gastric ulcer
* cancer
* uncontrolled bacterial, viral, fungal or parasite infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2016-09-28 (Actual); Primary Completion 2017-04-24 (Actual); Study Completion 2017-10-14 (Actual)

PRIMARY OUTCOMES:
Percent reduction in sum of the five GERD score from baseline. | One week after last OMT
  The five GERD variables recorded at baseline and one week after the last treatment were degrees of "Heartburn", "Chest pain", "Acid in mouth", "Epigastric pain" and "Thoracic pain", each recorded on a 10 cm VAS. The response variables were percent reduction in sum of the five GERD variables from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Stig E Larsen, PhD, Principal Investigator — Norwegian Univesity of Life Sciences

IPD SHARING:
Plan to Share IPD: Undecided